CLINICAL TRIAL: NCT01455584
Title: Phase Ⅰ Study to Determine the Maximum Tolerated Dose of HM781-36B Continuously Given in Patients With Advanced Solid Tumors and to Assess the Food Effect on Pharmacokinetic Profile
Brief Title: Clinical Trial to Determine the MTD of HM781-36B in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-PHI-102
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Solid Malignancies
Keywords: HM781-36B
MeSH Terms: interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM781-36B (Experimental): HM781-36B
  Interventions: Drug: HM781-36B tablets

INTERVENTIONS:
Drug: HM781-36B tablets — Q1X28D/4W for HM781-36B tablets
  Other Names: HM781-36B

SUMMARY:
The main objective of this study is to determine the maximum tolerated dose (MTD) of HM781-36B continuously.

DETAILED DESCRIPTION:
Besides the main objective, there are 4 other objectives as follows:

1. To determine dose-limiting toxicity (DLT) of HM781-36B
2. To determine Maximum Tolerated Dose (MTD) of HM781-36B
3. To determine the effect of food on the pharmacokinetics after dosed HM781-36B continuously
4. To evaluate anticancer activity of HM781-36B in patients with advanced solid malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced solid tumor
2. Patients who have experienced progressive disease despite of conventional anticancer therapy. Patients who cannot expect effective treatment or prolonged survival with conventional anticancer therapy
3. Previous chemotherapy, radiotherapy and surgical operation are allowed if they are discontinued for at least 4 weeks prior to D0 and all adverse events are resolved
4. Aged ≥19
5. Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2
6. A life expectancy greater than 12 weeks
7. Adequate bone marrow, renal and liver function.
8. Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up assessments and procedures

Exclusion Criteria:

1. Patients with hematopoietic malignancies,uncontrolled infection, CNS metastasis.
2. Patients who have undergone hematopoietic stem cell transplantation (HSCT) or are candidates for planned HSCT
3. Patients who have GI malabsorption or difficulty taking oral medication
4. Patients who have psychiatric or congenital disorder
5. Subjects who, in the investigator's opinion, cannot be treated per protocol due to functional impairments
6. Pregnant or breast-feeding patients; Women of childbearing potential without adequate contraception (Men must use adequate contraception.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
MTD determination | Dose limiting Toxicity will be evaluated on Day 28 during Cycle 1

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea